CLINICAL TRIAL: NCT03571815
Title: Cost Effectiveness of Sodium Fluoride Varnish Application in Prevention of Dental Caries in School Children Between Age of 6 and 7 Years
Brief Title: Cost Effectiveness of Sodium Fluoride Varnish in Prevention of Dental Caries in School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Peradeniya (Other)
Responsible Party: Principal Investigator, Dr. RM Jayasinghe, Principal investigator, University of Peradeniya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UPeradeniya
Record Dates: First submitted 2018-05-03; First posted 2018-06-28 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Dental Caries in Children
Keywords: Fluoride varnish; clinical trial; dental caries
MeSH Terms: conditions — Dental Caries | interventions — Bifluorid 12

STUDY DESIGN:
Masking Description: interventional group-fluoride varnish application. control group-water
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- fluoride varnish application (Experimental): intervention; fluoride varnish application (with 5% Sodium fluoride varnish application on teeth)
  Interventions: Drug: 5% sodium fluoride varnish
- control group (Placebo Comparator): application of water on teeth in the control group
  Interventions: Other: WATER ON TEETH

INTERVENTIONS:
Drug: 5% sodium fluoride varnish — application of sodium fluoride varnish on teeth
  Other Names: sodium fluoride varnish
  Arms: fluoride varnish application
Other: WATER ON TEETH — control group
  Arms: control group

SUMMARY:
Fluoride varnish application is universally accepted as a dental caries prevention method. This study was aimed in assessment of clinical outcome and cost effectiveness in using that method in Sri Lankan school children

DETAILED DESCRIPTION:
Background Dental caries remains a significant public health problem with multiple factors such as socioeconomic, dietary and microbiological playing a major role as risk factors in initiation and continuation of the disease. It is considered the most common cause of toothache and hospital admissions in young children. Dental caries in school children not only causes pain, but also affects school attendance, parents' work hours, children's ability to eat, play, rest and sleep. Therefore, dental caries when present significantly reduces the health related quality of life of a child.

Improving oral health has been considered as an objective in preventive dental care for children. Therefore the measures taken to prevent dental caries should include bacterial bio film control, dietary counseling, use of fluoride products such as toothpastes, mouth rinses, varnishes, gels and foams, and Casein phosphopeptide (CPP) - amorphous calcium phosphate (ACP) cream and gums and placing resin-based/glass ionomer pit and fissure sealants.) Professional fluoride varnish application has become popular among all methods as variety of studies has discussed its effect in reducing dental caries.

Fluoride varnish use in the U.S. has increased markedly since it was approved by the FDA in 1994. Fluoride varnish's effectiveness in caries prevention, ease of application, and safety give it an advantage over other types of topical fluoride treatments (such as gels and rinses) or other caries management methods. As a result, it is regarded as one of the superior topical fluoride agents for young children. Fluoride varnish also prolongs the contact time between fluoride and tooth surface to reduce caries. Its active ingredient is usually 5% sodium fluoride, or 22,600 ppm fluoride. It also has recently gained much attention in dentistry because the risk of dental fluorosis is found to be minimal.The simplicity of its application makes it very suitable and practical for use in different places and groups.

Justification Despite the availability of free health dental service in Sri Lanka, the prevalence and severity of dental caries among six and seven years old school children stand at a very high level according to the results of national oral health survey as 78% (83/84), 76.4% (94/95) and 65.5% (2002/2003) whereas the dmft is 4.4, 4.1 and 3.6.9 The simplicity of fluoride varnish application makes it very suitable and practical for use in dental clinics and outreach dental services, especially in young children and in other special needs groups.

Up to date to our knowledge, there was no other study carried out on cost effectiveness of fluoride varnish application on teeth in Sri Lankan population. Therefore, the results of the study will be beneficial in implementation and identification of advantages of fluoride varnish application on teeth in young children.

Aim The main objective of this study was to evaluate the cost effectiveness of six monthly application of sodium fluoride varnish in prevention of dental caries in deciduous teeth, permanent incisors and molars in children between six and seven years in Sri Lanka.

The specific objective is

1. To find out the association between dental caries and the social status of the child (e.g. mother's education, father's education, monthly family income etc.)

Methods Study Type: Interventional This was a double-blind, randomized controlled trial. A sample of school children (6-7 years) were randomized into varnish and control groups. All the children received routine caries preventive measures of oral hygiene instructions, dietary advice and professional cleaning. Children in fluoride varnish application group received fluoride varnish professionally applied after prophylaxis every 6 months combined with counseling on maintenance of oral hygiene and diet for a period of 2 years. Clinical examinations of all children were performed at the beginning of the study and 1 year and 2 years later. All the caries at the dentinal level of both groups were stabilized with temporary restorations at the beginning. For evaluation and comparison, all the collected data was subjected to statistical analysis. Both varnish and control groups were subjected to use of fluoride tooth paste of 1000ppm. The control group was subjected to counseling on maintenance of oral hygiene and diet. During this period, the team visited each school four times at six months interval for recruitment, dental examinations, and fluoride varnish applications. Recruited children were randomly assigned to either a treatment (5% Sodium Fluoride varnish) or a control group. Trained interviewers collected data on oral health habits and sociodemographic characteristics of the children. Information on the child's diet was collected through a 4-day food frequency diary. Caries examinations were conducted using the International Caries Detection and Assessment System (ICDAS). The cost for the dental team's school visits; cost involved in the treatment of dental caries throughout the course of the study in both groups were evaluated and compared at the end of the study.

The sample size was calculated as 160 each arm to detect 5% caries change with 80% power.

Analysis The effect of intervention was measured in terms of number of caries prevented. The number of new caries in the usual care and intervention group was calculated after the completion of the study. The demographic and socioeconomic data of the intervention and usual care group were collected. The costs for intervention were estimated. The cost of treatment for caries was estimated for intervention and non-Intervention groups. The costs for the dental material, time for human resources and indirect costs were also calculated. The results were presented as cost per caries prevented.

ELIGIBILITY:
Inclusion Criteria:

* Children with at least one permanent tooth present.
* Age 6 to 7 years. Children under 6 years of age were enrolled in the study if at least one permanent tooth has erupted.
* Residing in Kurunegala municipal council region and tap water is consumed (fluoride levels in drinking water is normal).
* Consent from parental/ primary caregiver/ legal guardian or a family member who is the primary care provider.

Exclusion Criteria:

* Children with ulcerative gingivitis and stomatitis. (These children were referred for treatment.)
* No permanent teeth present or stainless steel crowns only

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2015-01-02 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-07-02 (Actual)

PRIMARY OUTCOMES:
change of number of teeth with dental caries at 6months, 1 year and 2 years from the initial presentation | 2years
  change of number of new dental caries prevented using sodium fluoride varnish application at 6months, 1 year and 2years from the initial presentation for the study